CLINICAL TRIAL: NCT07265505
Title: Study of Immune and Microbiological Modifications of the Endometrium in Cases of Recurrent Implantation Failure and/or Recurrent Pregnancy Loss
Brief Title: Study of Endometrial Immune and Microbiological Modifications in Cases of Recurrent Implantation Failure and/or Recurrent Pregnancy Loss
Acronym: IMERR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); ADREGOF (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP241344; 2024-A02100-47 (Other: France : Ministry of Health)
Record Dates: First submitted 2025-05-26; First posted 2025-12-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Implantation Failure; Recurrent Pregnancy Loss; Infertility, Female; Endometrial Diseases; Endometritis; Endometriosis; Adenomyosis
Keywords: Uterine Immune Profile; Endometrial Receptivity; Infertility; Recurrent Miscarriage; IVF Failure; Implantation Window; Reproductive Immunology; Endometrial Microbiome; Chronic Endometritis; Adenomyosis; Endometriosis
MeSH Terms: conditions — Infertility, Female; Uterine Diseases; Endometritis; Endometriosis; Adenomyosis; Infertility; Abortion, Habitual | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIF/RPL group (Other): Women undergoing ART with a history of recurrent implantation failure (RIF) and/or recurrent pregnancy loss (RPL).
  Interventions: Diagnostic Test: Endometrial Biopsy; Diagnostic Test: Vaginal Swab; Diagnostic Test: Blood sample; Diagnostic Test: Pelvic ultrasound (±pelvic MRI)
- Control group (Other): Women undergoing ART without a history of RIF or RPL.
  Interventions: Diagnostic Test: Endometrial Biopsy; Diagnostic Test: Vaginal Swab; Diagnostic Test: Blood sample; Diagnostic Test: Pelvic ultrasound (±pelvic MRI)

INTERVENTIONS:
Diagnostic Test: Endometrial Biopsy — Endometrial biopsy with Cornier Pipelle (part of the treatment in the RIF/RPL group and some patients of the control group / added for the research for the other patients of the control group)
Diagnostic Test: Vaginal Swab — Vaginal sample collection using a cotton swab. Part of the treatment
Diagnostic Test: Blood sample — Peripheral blood draw. Part of the treatment + 10 mL additional for research
Diagnostic Test: Pelvic ultrasound (±pelvic MRI) — Pelvic ultrasound (±pelvic MRI). Part of the treatment

SUMMARY:
The IMERR study aims to improve understanding of certain causes of infertility related to recurrent implantation failure (RIF) and/or recurrent pregnancy loss (RPL), conditions that affect many women undergoing assisted reproductive technology (ART). Despite medical advances, some patients repeatedly fail to achieve pregnancy, or experience repeated miscarriages. These situations may be linked to subtle immune or microbial disturbances in the uterus. This study seeks to identify immune and microbiological profiles in the endometrium during the implantation window-a crucial period when the embryo attaches to the uterine wall. We will compare women who have experienced RIF and/or RPL with women who have had no such history. Blood and uterine samples will be analyzed to investigate whether certain immune or microbial features are associated with these reproductive failures. The ultimate goal is to uncover predictive factors that may explain why some women experience implantation failure or pregnancy loss, and to lay the foundation for future personalized treatments to improve reproductive outcomes.

DETAILED DESCRIPTION:
The IMERR study is a prospective, monocentric, controlled interventional study aiming to identify immune and microbiological signatures in the eutopic endometrium of women undergoing ART (IVF/ICSI), with and without a history of recurrent implantation failure (RIF) and/or recurrent pregnancy loss (RPL). RIF is defined as the absence of clinical pregnancy after at least three embryo transfers of good-quality blastocysts, and RPL as two or more consecutive pregnancy losses before 24 weeks of gestation.

Participants will be divided into two groups: a study group (with RIF and/or RPL) and a control group (without RIF or RPL). Endometrial biopsies will be collected during the implantation window, alongside peripheral blood and vaginal samples. These samples will undergo immunological and microbiological analyses, including histology, immunophenotyping, and microbiota profiling.

The study aims to (i) Characterize immune cell populations in the endometrium and blood, (ii) Investigate the endometrial microbiome and its potential dysbiosis, (iii) Explore associations between these biological profiles and clinical features such as endometriosis, adenomyosis, chronic endometritis, or uterine contractility disorders.

The study includes 100 participants and spans a total duration of 60 months (36 months for inclusion and 24 months of follow-up). A subgroup analysis will assess the association between immuno-microbiological profiles and clinical outcomes after embryo transfer within the 24-month post-inclusion period.

By identifying predictive markers of RIF and RPL, this study may help establish new diagnostic tools and personalized treatment strategies in reproductive medicine.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥18 and <36 years
* Undergoing assisted reproductive technology (ART) in a fertility center
* Covered by the French national health insurance system
* Belonging to one of two groups:

  * Study group: history of recurrent implantation failure (RIF) and/or recurrent pregnancy loss (RPL)
  * Control group: no history of RIF or RPL

Exclusion Criteria:

* Pregnant at inclusion
* Refusal to provide written informed consent
* Antibiotic use within one month prior to endometrial biopsy Positive serology for hepatitis B, hepatitis C or HIV
* Uterine anatomical abnormalities (e.g., polyps, cavity-distorting fibroids, untreated hydrosalpinx)
* Known chromosomal abnormality in either partner
* Known autoimmune disease, thrombophilia, or antiphospholipid antibody syndrome
* Persons under legal protection (e.g., guardianship, curatorship)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Profiling of endometrial immune cell populations | Baseline
  Profiling of endometrial immune cell populations (proportion of subpopulation) during the implantation window using single-cell transcriptomics and/or flow cytometry.
  Endometrial biopsies will be collected during the implantation window. Immune cell populations will be characterized using either single-cell RNA sequencing (scRNA-seq) and /or multiparametric flow cytometry, depending on technical feasibility and sample quality. For scRNA-seq, transcriptomic analysis will be performed (e.g., using the 10x Genomics platform), and immune cell types will be identified via clustering and annotation algorithms. For flow cytometry, immune subsets will be identified and quantified based on surface marker expression. Comparisons of immune profiles will be made between women with and without a history of RIF and/or RPL.

SECONDARY OUTCOMES:
Microbiological profiling of endometrial tissue | Baseline
  Microbiological profiling of endometrial tissue during the implantation window using next-generation sequencing (NGS)
  Endometrial microbiota will be characterized by next-generation sequencing (NGS) of DNA extracted from endometrial biopsy samples collected during the implantation window. Diversity metrics (alpha and beta diversity) and relative abundances of microbial taxa will be compared between women with and without a history of RIF and/or RPL.
Characterization of peripheral blood immune cell populations | Baseline
  Characterization of peripheral blood immune cell populations during the implantation window using single-cell transcriptomics and/or flow cytometry
  Peripheral blood samples will be collected at inclusion. Immune profiling will be performed to characterize circulating immune cell subpopulations. Depending on feasibility and sample quality, either single-cell RNA sequencing (scRNA-seq) and / or multiparametric flow cytometry may be used. Immune profiles will be compared between women with and without a history of RIF and/or RPL.
Exploratory analysis of associations between immune and microbiological profiles and clinical, radiological, and histological characteristics | Baseline
  This outcome consists of exploratory analyses assessing the associations between previously measured immune and microbiological profiles (from endometrial tissue) and (i) clinical outcomes (e.g., pregnancy, miscarriage, live birth), (ii) radiological findings (e.g., adenomyosis, uterine contractility), and (iii) histological/bacteriological findings (e.g., chronic endometritis with CD138+ cells or vaginal cultures). No new biological measurements will be performed. Each association will be reported as a separate statistical outcome (e.g., odds ratios, p-values)
Exploratory analysis of associations between immune and microbiological profiles and clinical, radiological, and histological characteristics | Through 24 months of follow-up
  This outcome consists of exploratory analyses assessing the associations between previously measured immune and microbiological profiles (from endometrial tissue) and (i) clinical outcomes (e.g., pregnancy, miscarriage, live birth), (ii) radiological findings (e.g., adenomyosis, uterine contractility), and (iii) histological/bacteriological findings (e.g., chronic endometritis with CD138+ cells or vaginal cultures). No new biological measurements will be performed. Each association will be reported as a separate statistical outcome (e.g., odds ratios, p-values)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Bourdon, MD, PhD, Principal Investigator — Service de Gynécologie Obstétrique II et Médecine de la Reproduction - Cochin Hospital
Locations (1):
- Service de Gynécologie Obstétrique II et Médecine de la Reproduction - Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benner M, Ferwerda G, Joosten I, van der Molen RG. How uterine microbiota might be responsible for a receptive, fertile endometrium. Hum Reprod Update. 2018 Jul 1;24(4):393-415. doi: 10.1093/humupd/dmy012. PMID 29668899
- [Background] Bourdon M, Santulli P, Jeljeli M, Vannuccini S, Marcellin L, Doridot L, Petraglia F, Batteux F, Chapron C. Immunological changes associated with adenomyosis: a systematic review. Hum Reprod Update. 2021 Jan 4;27(1):108-129. doi: 10.1093/humupd/dmaa038. PMID 33099635
- [Background] Campo S, Campo V, Benagiano G. Infertility and adenomyosis. Obstet Gynecol Int. 2012;2012:786132. doi: 10.1155/2012/786132. Epub 2011 Dec 26. PMID 22242025
- [Background] Chen P, Chen P, Guo Y, Fang C, Li T. Interaction Between Chronic Endometritis Caused Endometrial Microbiota Disorder and Endometrial Immune Environment Change in Recurrent Implantation Failure. Front Immunol. 2021 Oct 4;12:748447. doi: 10.3389/fimmu.2021.748447. eCollection 2021. PMID 34671363
- [Background] Duffy JMN, Adamson GD, Benson E, Bhattacharya S, Bhattacharya S, Bofill M, Brian K, Collura B, Curtis C, Evers JLH, Farquharson RG, Fincham A, Franik S, Giudice LC, Glanville E, Hickey M, Horne AW, Hull ML, Johnson NP, Jordan V, Khalaf Y, Knijnenburg JML, Legro RS, Lensen S, MacKenzie J, Mavrelos D, Mol BW, Morbeck DE, Nagels H, Ng EHY, Niederberger C, Otter AS, Puscasiu L, Rautakallio-Hokkanen S, Sadler L, Sarris I, Showell M, Stewart J, Strandell A, Strawbridge C, Vail A, van Wely M, Vercoe M, Vuong NL, Wang AY, Wang R, Wilkinson J, Wong K, Wong TY, Farquhar CM; Priority Setting Partnership for Infertility. Top 10 priorities for future infertility research: an international consensus development study. Fertil Steril. 2021 Jan;115(1):180-190. doi: 10.1016/j.fertnstert.2020.11.014. Epub 2020 Nov 30. PMID 33272617
- [Background] ESHRE Guideline Group on RPL; Bender Atik R, Christiansen OB, Elson J, Kolte AM, Lewis S, Middeldorp S, Mcheik S, Peramo B, Quenby S, Nielsen HS, van der Hoorn ML, Vermeulen N, Goddijn M. ESHRE guideline: recurrent pregnancy loss: an update in 2022. Hum Reprod Open. 2023 Mar 2;2023(1):hoad002. doi: 10.1093/hropen/hoad002. eCollection 2023. PMID 36873081
- [Background] ESHRE Working Group on Recurrent Implantation Failure; Cimadomo D, de Los Santos MJ, Griesinger G, Lainas G, Le Clef N, McLernon DJ, Montjean D, Toth B, Vermeulen N, Macklon N. ESHRE good practice recommendations on recurrent implantation failure. Hum Reprod Open. 2023 Jun 15;2023(3):hoad023. doi: 10.1093/hropen/hoad023. eCollection 2023. PMID 37332387
- [Background] Giuliani E, Parkin KL, Lessey BA, Young SL, Fazleabas AT. Characterization of uterine NK cells in women with infertility or recurrent pregnancy loss and associated endometriosis. Am J Reprod Immunol. 2014 Sep;72(3):262-9. doi: 10.1111/aji.12259. Epub 2014 May 8. PMID 24807109
- [Background] Kunz G, Leyendecker G. Uterine peristaltic activity during the menstrual cycle: characterization, regulation, function and dysfunction. Reprod Biomed Online. 2002;4 Suppl 3:5-9. doi: 10.1016/s1472-6483(12)60108-4. PMID 12470555
- [Background] Ledee N, Petitbarat M, Prat-Ellenberg L, Dray G, Cassuto GN, Chevrier L, Kazhalawi A, Vezmar K, Chaouat G. The uterine immune profile: A method for individualizing the management of women who have failed to implant an embryo after IVF/ICSI. J Reprod Immunol. 2020 Nov;142:103207. doi: 10.1016/j.jri.2020.103207. Epub 2020 Sep 14. PMID 32971456
- [Background] Marron K, Harrity C. Endometrial lymphocyte concentrations in adverse reproductive outcome populations. J Assist Reprod Genet. 2019 May;36(5):837-846. doi: 10.1007/s10815-019-01427-8. Epub 2019 Mar 7. PMID 30847699
- [Background] McQueen DB, Bernardi LA, Stephenson MD. Chronic endometritis in women with recurrent early pregnancy loss and/or fetal demise. Fertil Steril. 2014 Apr;101(4):1026-30. doi: 10.1016/j.fertnstert.2013.12.031. Epub 2014 Jan 23. PMID 24462055
- [Background] Ota H, Tanaka T. Stromal vascularization in the endometrium during adenomyosis. Microsc Res Tech. 2003 Mar 1;60(4):445-9. doi: 10.1002/jemt.10282. PMID 12567401
- [Background] Pirtea P, Cicinelli E, De Nola R, de Ziegler D, Ayoubi JM. Endometrial causes of recurrent pregnancy losses: endometriosis, adenomyosis, and chronic endometritis. Fertil Steril. 2021 Mar;115(3):546-560. doi: 10.1016/j.fertnstert.2020.12.010. Epub 2021 Feb 11. PMID 33581856
- [Background] Rimmer MP, Fishwick K, Henderson I, Chinn D, Al Wattar BH, Quenby S. Quantifying CD138+ cells in the endometrium to assess chronic endometritis in women at risk of recurrent pregnancy loss: A prospective cohort study and rapid review. J Obstet Gynaecol Res. 2021 Feb;47(2):689-697. doi: 10.1111/jog.14585. Epub 2020 Dec 3. PMID 33274569
- [Background] Romero R, Espinoza J, Mazor M. Can endometrial infection/inflammation explain implantation failure, spontaneous abortion, and preterm birth after in vitro fertilization? Fertil Steril. 2004 Oct;82(4):799-804. doi: 10.1016/j.fertnstert.2004.05.076. PMID 15482749
- [Background] Vernon M, Stern JE, Ball GD, Wininger D, Mayer J, Racowsky C. Utility of the national embryo morphology data collection by the Society for Assisted Reproductive Technologies (SART): correlation between day-3 morphology grade and live-birth outcome. Fertil Steril. 2011 Jun 30;95(8):2761-3. doi: 10.1016/j.fertnstert.2011.02.008. Epub 2011 Mar 15. PMID 21406305
- [Background] Von Woon E, Greer O, Shah N, Nikolaou D, Johnson M, Male V. Number and function of uterine natural killer cells in recurrent miscarriage and implantation failure: a systematic review and meta-analysis. Hum Reprod Update. 2022 Jun 30;28(4):548-582. doi: 10.1093/humupd/dmac006. PMID 35265977
- [Background] Zhao Y, Chen X, Zhang T, Chan LKY, Liu Y, Chung JP, Kwong J, Li TC. The use of multiplex staining to measure the density and clustering of four endometrial immune cells around the implantation period in women with recurrent miscarriage: comparison with fertile controls. J Mol Histol. 2020 Oct;51(5):593-603. doi: 10.1007/s10735-020-09908-2. Epub 2020 Aug 28. PMID 32857228